CLINICAL TRIAL: NCT05713773
Title: Pharmacodynamics and Pharmacokinetics of 3 New Developed Coated Glucose Beads Formulations After Single-dose Administration (Fasting Conditions) in 20 Obese Healthy Subjects
Brief Title: Pharmacodynamics and Pharmacokinetics of 3 New Developed Coated Glucose Beads in 20 Obese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aphaia Pharma US LLC (Industry)
Collaborators: ACC GmbH Analytical Clinical Concepts, Germany (Unknown); Nova-Clin Medical Research Center S.R.L., Romania (Unknown); BioClinica, Inc. (Industry); Galephar Pharmaceutical Research (PR), Inc, Puerto Rico (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 017B19
Record Dates: First submitted 2023-01-19; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Intervention Model Description: single-dose, randomized, open label, five-treatment, five-period, five-sequence crossover, at one study site
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Test product 1 (T1) (Active Comparator): Aphaia Pharma (APH)-001A: glucose coated beads containing 8 g glucose and caffeine anhydrous
  Interventions: Drug: coated beads glucose (8 g) and caffeine anhydrous
- Test product 2 (T2) (Active Comparator): APH-001B: glucose coated beads containing 8 g glucose and caffeine anhydrous
  Interventions: Drug: coated beads glucose (8 g) and caffeine anhydrous
- Test product 3 (T3) (Active Comparator): APH-001C: glucose coated beads containing 8 g glucose and caffeine anhydrous
  Interventions: Drug: coated beads glucose (8 g) and caffeine anhydrous
- Test product 4 (T4) (Active Comparator): APH-001D: glucose coated beads containing 8 g glucose
  Interventions: Drug: coated beads glucose (8 g)
- Test product 5 (T5) (Active Comparator): APH-001E: uncoated beads containing 8 g glucose and caffeine anhydrous
  Interventions: Drug: uncoated beads glucose (8 g) and caffeine anhydrous

INTERVENTIONS:
Drug: coated beads glucose (8 g) and caffeine anhydrous — After an overnight fasting of about 10 hours the subjects were administered either glucose (8 g) or glucose (8 g) and caffeine starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position on Day 1.
  Other Names: APH-001A
  Arms: Test product 1 (T1)
Drug: coated beads glucose (8 g) and caffeine anhydrous — After an overnight fasting of about 10 hours the subjects were administered either glucose (8 g) or glucose (8 g) and caffeine starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position on Day 1.
  Other Names: APH-001B
  Arms: Test product 2 (T2)
Drug: coated beads glucose (8 g) and caffeine anhydrous — After an overnight fasting of about 10 hours the subjects were administered either glucose (8 g) or glucose (8 g) and caffeine starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position on Day 1.
  Other Names: APH-001C
  Arms: Test product 3 (T3)
Drug: coated beads glucose (8 g) — After an overnight fasting of about 10 hours the subjects were administered glucose (8 g) starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position on Day 1.
  Other Names: APH-001D
  Arms: Test product 4 (T4)
Drug: uncoated beads glucose (8 g) and caffeine anhydrous — After an overnight fasting of about 10 hours the subjects were administered either glucose (8 g) or glucose (8 g) and caffeine starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position on Day 1.
  Other Names: APH-001E
  Arms: Test product 5 (T5)

SUMMARY:
This single-dose, randomized, open label, five-treatment, five-period, five-sequence crossover study was performed to assess pharmacodynamics (PD) and pharmacokinetics (PK) of three new developed coated Glucose beads formulations (containing glucose (8 g) and caffeine), one coated Glucose beads formulation (containing glucose (8 g)) and one uncoated Glucose beads formulation (containing Glucose (8 g) and caffeine) after single-dose administration (fasting conditions) in 20 obese healthy subjects. After an overnight fasting of at least 10 hours the subjects were administered either glucose (8 g) or glucose (8 g) and caffeine starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position. At least 3 days wash-out period was kept between each treatment periods.

DETAILED DESCRIPTION:
This single-dose, randomized, open label, five-treatment, five-period, five-sequence crossover study was performed to assess pharmacodynamics (PD) and pharmacokinetics (PK) of three new developed coated Glucose beads formulations (containing glucose (8 g) and caffeine), one coated Glucose beads formulation (containing glucose (8 g)) and one uncoated Glucose beads formulation (containing Glucose (8 g) and caffeine) after single-dose administration (fasting conditions) in 20 obese healthy subjects.

Only subjects who had given voluntarily their informed consent participated in the screening examination and, if found eligible as per study inclusion and exclusion criteria, were enrolled in the study. At least 13 hours before investigational product administration in each treatment period, subjects were admitted to the clinical site. During each treatment period the hospitalization period in the clinical unit was 13 hours before and up to 11 hours after investigational product administration.

Test products (T1, T 2, T3, T4, T5) was administered as single oral doses during the first, second, third, fourth and fifth treatment period corresponding to the randomization code under fasting conditions.

After an overnight fasting of at least 10 hours, the subjects were administered either glucose (8 g) or glucose (8 g) and caffeine starting at 8:00 (time 0; administration time was staggered beginning at 8:00 for the first group of subjects) in sitting position. According to the randomization code subjects were received on the respective study day one coated beads formulations (T1, T2, T3, T 4) or the uncoated beads formulation (T5).

A total of 17 blood samples were drawn for determination of Glucagon-like peptide-1 (GLP-1) levels and pharmacokinetic analysis of caffeine at the prescribed times, pre-dose (1.0 h, 0.5 hand 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration. Blood samples for glucose measurements was taken via an indwelling catheter or vein puncture from the forearm vein pre-dose (1.0 h, and 0 h) and at 0.5, 1.0, 2.0, 3.0, 4 0, 5.0, 6 0, 8.0 and 10.0 hours after investigational product administration.

Visual analogue scale (VAS) (appetite), VAS (stomach rumbles) were evaluated at the prescribed times pre-dose (0 h) and at 2, 4 and 10 hours after investigational product administration.

Wash-out periods of at least 3 days were separated the five treatment periods.

Within 7 days after last blood sampling in the last treatment period 12-lead electrocardiogram (ECG), vital signs, clinical routine laboratory parameters, physical examination and check of adverse events were repeated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy obese, Caucasian male and female subjects 18 - 55 years of age
* Body mass index within the range of > 30.0 kg/m2
* Waist circumference: men > 102 cm; women > 88 cm
* Female subjects of childbearing potential agree to undergo pregnancy tests and to use an appropriate method of contraception (i.e., oral contraceptive steroids, intrauterine device, barrier method)
* Findings within the range of clinical acceptability in medical history (or the clinical investigator considers the deviation to be irrelevant for the purpose of the study)
* Findings within the range of clinical acceptability in physical examination (or the clinical investigator considers the deviation to be irrelevant for the purpose of the study)
* Laboratory values within the normal range (or the clinical investigator considers the deviation to be irrelevant for the purpose of the study)
* Normal ECG or abnormalities which the clinical investigator does not consider a disqualification for participation in the study
* Normal vital signs (normal blood pressure and heart rate measured under stabilized conditions at screening visit after at least 5 minutes of rest in sitting position) or abnormalities which the clinical investigator does not consider a disqualification for participation in the study
* Normal gastrointestinal (GI) function or abnormalities which the clinical investigator does not consider a disqualification for participation in the study
* Willingness to undergo screening and follow-up examinations (i.e., physical examinations and laboratory investigations before and after the treatment periods)
* Ability to comprehend subject information and willingness to sign the informed consent
* Non-smokers or mild to moderate smokers (less or equal 10 cigarettes daily)

Exclusion Criteria:

* Gastrointestinal, hepatic and renal diseases and/or pathological findings which might interfere with pharmacokinetics and pharmacodynamics of the investigational product
* Established diagnosis of type-1 or type-2 diabetes mellitus
* Treatment with insulin, insulin secretagogues (sulfonylurea derivatives, glinides, GLP-1 agonists (exenatide, lixisenatide, glutides), or thiazolidinediones (glitazones)
* Unexplained rise in blood glucose
* Treatment for constipation (including but not limited to lactulose or any other form of stool softeners, laxatives) or diarrhea (including but not limited to pectins. loperamide etc.) or any other medication known to interfere with gastrointestinal transit time, such as e.g., metoclopramide, opioids, or gastric Potential of Hydrogen (pH) (including but not limited to antacids, H2-receptor antagonists, prazole)
* Tea, coffee or other caffeine containing beverage drinkers (more than 0.4 L per day)
* History of hypersensitivity to the investigational product or any related drugs or to any of the excipients
* History or presence of any clinically significant cardiovascular, pulmonary, hepatobiliary, renal, hematological, gastrointestinal, endocrinologic, immunologic, dermatologic. neurological, psychiatric, metabolic, musculoskeletal, or malignant disease, which the clinical investigator does not consider a disqualification for participation in the study
* Known heart failure (Grade I to IV of New York Heart Association classification)
* Significant renal disease. including nephritic syndrome chronic renal failure (defined as creatinine clearance< 60 mL/min and serum creatinine >180 μmol/L)
* Unexplained serum creatine phosphokinase (CPK) > 3-times the upper limit of normal (ULN) Subjects with a reason for CPK elevation may have the measurement repeated prior to randomization a CPK retest> 3-times ULN leads to exclusion
* Clinically significant illness or surgery within 4 weeks prior to dosing
* Less than 14 days after last acute disease
* Volunteers liable to orthostatic dysregulation, fainting, or blackouts
* Donation or loss of blood equal to or exceeding 500 ml during 90 days before the first administration of investigational product
* Participation in another study with an experimental drug within at least 3 months (or within five elimination half-lives of the previous experimental drug, whichever is longer) before the first administration of investigational product
* Any use of drug, prescribed or over-the-counter (OTC) (inclusive herbal remedies), within 2 weeks (or within six elimination half-lives of this medication, whichever is longer) prior to the first administration of investigational product except if this will not affect the outcome of the study in the opinion of the clinical investigator
* Unwillingness or inability to comply with the study protocol or study-related procedures (e.g., difficulty to stay fasting, consume the standard meals, or swallow the beads formulations; difficult venous access).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
GLP-1 | Pre-dose (-1.0 h, -0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  Area under the plasma concentration-time curve (AUC(0-t))
GLP-1 | Pre-dose (-1.0 h, -0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  AUC(1.5h-6h)
GLP-1 | Pre-dose (-1.0 h, -0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  Adjusted area under the plasma concentration-time cur (AUCadj(1.5h-6h))
GLP-1 | Pre-dose (-1.0 h, -0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  Maximum plasma concentration (Cmax(0-t))
GLP-1 | Pre-dose (-1.0 h, -0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  Cmax(1.5h-6h)
GLP-1 | Pre-dose (-1.0 h, -0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  Cmax,adj(1.5h-6h)
GLP-1 | Pre-dose (-1.0 h, -0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  time to reach maximum plasma concentration (tmax(0-t))
GLP-1 | Pre-dose (-1.0 h, -0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  tmax(1.5h-6h)
GLP-1 | Pre-dose (-1.0 h, -0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  Duration of time during the concentration in the plasma concentration-time curve exceeds at least 50 % of Cmax(1.5h-6h)

SECONDARY OUTCOMES:
Pharmacokinetics of Caffeine | Pre-dose (1.0 h, 0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  AUC(0-t)
Pharmacokinetics of Caffeine | Pre-dose (1.0 h, 0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  Cmax(0-t)
Pharmacokinetics of Caffeine | Pre-dose (1.0 h, 0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  tmax(0-t)
Pharmacokinetics of Caffeine | Pre-dose (1.0 h, 0.5 h and 0 h) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 8.0 and 10.0 hours after investigational product administration
  tlag
Pharmacokinetics of Glucose | Venous blood glucose measurement at the prescribed times pre-dose (-1.0 h, 0 h) and 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0 and 10.0 hours after investigational product administration
  AUC(0-t)
Pharmacokinetics of Glucose | Venous blood glucose measurement at the prescribed times pre-dose (-1.0 h, 0 h) and 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0 and 10.0 hours after investigational product administration
  Cmax(0-t)
Pharmacokinetics of Glucose | Venous blood glucose measurement at the prescribed times pre-dose (-1.0 h, 0 h) and 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0 and 10.0 hours after investigational product administration
  tmax(0-t)
Visual analogue scale (VAS) appetite | VAS (appetite) at the prescribed times pre-dose (0 h) and 2, 4 and 10 hours after investigational product administration.
  VAS for appetite with score of 1 - 10 was measured
VAS stomach rumbles | VAS (stomach rumbles) at the prescribed times pre-dose (0 h) and 2, 4 and 10 hours after investigational product administration.
  VAS for stomach rumbles with score of 1 - 10 was measured
Tolerability and safety | Within 7 days after last blood sampling in the last treatment period
  12-lead ECG
Tolerability and safety | Within 7 days after last blood sampling in the last treatment period
  vital signs
Tolerability and safety | Within 7 days after last blood sampling in the last treatment period
  clinical routine laboratory parameters
Tolerability and safety | Within 7 days after last blood sampling in the last treatment period
  physical examination
Tolerability and safety | Within 7 days after last blood sampling in the last treatment period
  check of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Vizman, Doctor, Principal Investigator — Aphaia Pharma AG
Locations (1):
- Nova-Clin Medical Research Center S.R.L.,, Timișoara, Romania

IPD SHARING:
Plan to Share IPD: No